CLINICAL TRIAL: NCT06699563
Title: The Effect of Using Motivational Cards on Pain Level and Number of Steps in Mobilization of Patients After Open Prostate Surgery
Brief Title: The Effect of Using a Motivation Card on Pain and Number of Walking Steps After Prostate Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Seher Ünver, Associate Professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/442
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Prostatic Hyperplasia
Keywords: Walking; Pain; Motivation
MeSH Terms: conditions — Prostatic Hyperplasia; Pain

STUDY DESIGN:
Intervention Model Description: The research will be conducted using randomized controlled, experimental type and single-blind research methods. For this purpose, after the data are collected, they will be coded as A and B groups, so the researcher who will make the research statistics will analyze the data without knowing the study and control groups. Randomization method will be used to determine the groups. For this, the patients who meet the study criteria and volunteer will be assigned to the groups using the randomization program 'Random Allocation Software 2.0' according to the order of hospitalization.
Masking Description: The data analyse is going to be completed by a independent researcher.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Experimental (with Card) (Experimental): In this procedure, patients used a pedometer and mobilization motivation card during their mobilization on the first postoperative day.
  Interventions: Behavioral: Mobilization Motivation Card
- No Intervention: Standard (No Card) (No Intervention): In this procedure, patients used a pedometer during their mobilization on the first postoperative day. They did not use a mobilization motivation card.

INTERVENTIONS:
Behavioral: Mobilization Motivation Card — On the morning of the surgery, the Mobilization Motivation Card and Pedometer will be introduced and the patient will be informed. On the morning of the first postoperative day, before the patient's first mobilization, pain assessment will be made with the Visual Analog Scale (VAS), and the Mobilization Motivation Card will be hung at the bedside during the day and will help increase the patient's participation in mobilization. Later, after a pedometer is attached to the patient's waist, the patient will be mobilized.
  Arms: Experimental: Experimental (with Card)

SUMMARY:
The purpose of this clinical study is to evaluate the effect of using motivational cards on pain and step counts in patients who underwent open prostate surgery due to benign prostatic hyperplasia.The main hypotheses are:

H1: Patients who use motivation cards during mobilization after open prostate surgery have lower pain levels than those who do not. H2: Patients who used motivation cards for mobilization after open prostate surgery had a higher number of steps than those who did not use them. After the surgery, patients were asked to walk with a pedometer. A mobilization motivation card was used in the study group.

DETAILED DESCRIPTION:
The group distribution of the patients was made using the Random Allocation Software (Version 2.0.0) program and the patients were divided into two groups: the study group and the control group.

The patients were visited by the researcher in their rooms on the morning of the day they were scheduled for surgery, and the purpose of the study was explained to the patients. Verbal and written consent was obtained from those who agreed to participate in the study, and it was explained to the patients that they would be visited again at their bedsides the day after surgery.

The Visual Pain Scale was created to assess the severity of pain. A score of '0' at the left end of the line indicates no pain, and a score of '10' at the right end indicates unbearable pain. In this study, patients were asked to mark the severity of the pain they were experiencing on a scale. The research nurse visited the patient in the service rooms before they were transferred to the operating room to make the first assessment in the study group, and the purpose of the study was explained to the patient. Patient introduction form, pedometer and mobilization motivation card were introduced to the patient. The patient was informed that they would be visited at 10:00 a.m. on the first day after the surgery to mobilize the patient. On the morning of the first day after surgery, the patient's pain status was determined with the Visual Pain Scale. The patient's vital signs were checked and the pedometer was placed on the lumbar region. The patient was mobilized according to the mobilization stage. The number of steps after the first mobilization was recorded on the mobilization motivation card and the card was hung at the bedside. The researcher nurse was informed that he would be visited again in 1 hour and these stages were repeated 3 times.

In the control group, the first evaluation was made by the researcher nurse. Patient introduction form, pedometer were introduced to the patient. On the morning of the first day after surgery, the patient's pain status was determined with the Visual Pain Scale. The patient's vital signs were checked and the pedometer was placed on the lumbar region. The patient was mobilized according to the mobilization stage. The number of steps after the first mobilization was recorded on the mobilization motivation card but was not given to the patient. The researcher nurse informed that he would be visited again in 1 hour and these stages were repeated 3 times.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in the ENT-Urology Clinic
* Those aged 18 and over
* Those who will undergo elective surgery
* Volunteer to participate in the study
* Post-surgical follow-up will be done in the service.
* Those who will undergo general anesthesia
* No mental problems
* Patients who had no vision, hearing or speech problems were included.

Exclusion Criteria:

* Those who will undergo emergency and unplanned surgical intervention
* Laparoscopic surgery was performed
* Taken to the intensive care unit after surgery
* Those who will not undergo general anesthesia
* Having mental problems
* Patients with vision, hearing and speech problems were not included.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Number of steps after surgery | 12 months
  Before mobilization, the number of steps taken will be tracked via a pedometer placed on the patient's waist, and after mobilization, the pedometer will be taken back from the patient. The number of steps taken will be recorded by the nurse.

SECONDARY OUTCOMES:
Pain before and after mobilization | 12 months
  Before mobilization, patients will be assessed for pain using a visual analog pain scale. To assess pain, patients are asked to rate their pain level on a scale ranging from 0 - "No pain" to 10 - "Unbearable pain".

CONTACTS AND LOCATIONS:
Overall Officials: Seher Unver, Principal Investigator — Trakya University
Locations (1):
- Tekirdağ Dr. İsmail Fehmi Cumalıoğlu City Hospital, Tekirdağ, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No